CLINICAL TRIAL: NCT02910700
Title: A Phase II Study of the TRIplet Combination of Dabrafenib, Nivolumab, and Trametinib in Patients With Metastatic Melanoma (TRIDeNT) or Binimetinib, EnCorafenib, and NivolumAb (TRIBECA)
Brief Title: Nivolumab With Trametinib and Dabrafenib, or Encorafenib and Binimetinib in Treating Patients With BRAF Mutated Metastatic or Unresectable Stage III-IV Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0605; NCI-2016-01940 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0605 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Melanoma; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Unresectable Melanoma
MeSH Terms: conditions — Brain Neoplasms; Melanoma | interventions — binimetinib; dabrafenib; encorafenib; Nivolumab; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (NDT, CLOSED) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1, dabrafenib PO BID on days 1-28, and trametinib PO QD on days 1-28. Cycles repeats every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dabrafenib; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacological Study; Drug: Trametinib
- Arm B (NT, closed to accrual) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 and 15, and trametinib PO QD on days 1-28. Cycles repeats every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacological Study; Drug: Trametinib
- Arm C (NEB) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 and 15, encorafenib PO QD on days 1-28, and binimetinib PO BID on days 1-28. Cycles repeats every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Drug: Encorafenib; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacological Study

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Arms: Arm C (NEB)
Drug: Dabrafenib — Given PO
  Arms: Arm A (NDT, CLOSED)
Drug: Encorafenib — Given PO
  Arms: Arm C (NEB)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
Other: Pharmacological Study — Correlative studies
Drug: Trametinib — Given PO
  Arms: Arm A (NDT, CLOSED); Arm B (NT, closed to accrual)

SUMMARY:
This phase II trial studies the side effects and how well nivolumab with trametinib and dabrafenib, or encorafenib and binimetinib work in treating patients with BRAF-mutated stage III-IV melanoma that has spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Immunotherapy with monoclonal antibodies, such as nivolumab, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. Trametinib, dabrafenib, encorafenib, and binimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known if nivolumab with trametinib and dabrafenib, or encorafenib and binimetinib may work better in treating patients with BRAF-mutated melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, tolerability, and efficacy (objective response rates by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) of nivolumab in combination with dabrafenib and trametinib or encorafenib and binimetinib in patients with BRAF-mutated metastatic melanoma.

SECONDARY OBJECTIVES:

I. Safety and tolerability of the nivolumab, dabrafenib, and trametinib triplet combination (NDT).

II. Safety and tolerability of the nivolumab, binimetinib and encorafenib. III. Efficacy of the combination as measured by the depth and duration of response by RECIST 1.1 and modified RECIST 1.1 (to include intracranial response).

IV. Pharmacodynamic evaluation of combination on circulating markers (immune monitoring).

V. Pharmacodynamic evaluation of combination on tumor tissues. VI. Progression- free survival and overall survival.

OUTLINE: Patients are assigned to 1 of 3 arms.

ARM A (NDT, CLOSED): Patients receive nivolumab intravenously (IV) over 30 minutes on day 1, dabrafenib orally (PO) twice daily (BID) on days 1-28, and trametinib PO once daily (QD) on days 1-28. Cycles repeats every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.

ARM B (NT, CLOSED TO ACCRUAL): Patients receive nivolumab IV over 30 minutes on day 1 and 15, and trametinib PO QD on days 1-28. Cycles repeats every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.

ARM C (NEB): Patients receive nivolumab IV over 30 minutes on day 1 and 15, encorafenib PO QD on days 1-28, and binimetinib PO BID on days 1-28. Cycles repeats every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days then every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic melanoma (stage IV) or unresectable Stage III that have progressed on or after receiving prior PD-1 directed therapy; only patients with BRAF V600 mutated melanoma are eligible; please note that patients with brain metastasis are not required to have prior PD-1
* Prior therapies for metastatic melanoma are allowed, including chemo-, cytokine-, immuno, biological and vaccine-therapy as long as they did not include BRAFi, MEKi; patients who have progressed on or after receiving anti-PD-1therapy in the adjuvant setting are also allowed; prior ipilimumab and/or PD-1 directed therapy will be allowed with a washout period of 2 weeks and if all autoimmune adverse events have resolved to grade 1 (except endocrine abnormalities that require continuous replacement)
* Evidence of evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients with melanoma brain metastases are allowed regardless of prior PD-1 exposure. Subjects with brain metastases are eligible if:

  * Metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for 2 weeks after treatment is complete and within 14 days of the first dose of nivolumab administration; or
  * If they are untreated but asymptomatic; or
  * If they are untreated and symptomatic but symptoms are controlled on stable or decreasing doses of steroids for 14 days prior to drug administration; or
  * If they have untreated leptomeningeal disease (LMD) as long as they fulfill all other eligibility requirements.
  * Note: Patients are excluded if they require high doses of systemic corticosteroids (> 8 mg equivalent of dexamethasone) to control central nervous system (CNS) symptoms.
* White blood cells (WBC) >= 2000 /uL (within one week prior to registration)
* Neutrophils >= 1500 /uL (within one week prior to registration)
* Platelets >= 100 x 10^3 /uL (within one week prior to registration)
* Hemoglobin > 9.0 g/dL (within one week prior to registration)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) >= 40 mL/min (if using the Cockcroft-Gault formula) (within one week prior to registration)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN (within one week prior to registration)
* Total bilirubin =< 1.5 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL) (within one week prior to registration)
* Women of childbearing potential (WOCBP) must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug; WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the start of nivolumab
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) and azoospermic men do not require contraception
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients that had grade 3/4 immune-related adverse events (AEs) on ipilimumab or nivolumab that required more than 12 weeks of immune suppression with corticosteroids
* History of interstitial lung disease or pneumonitis
* History of known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Active, known or suspected autoimmune disease; subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism and/or hypophysitis due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Require systemic treatment with either corticosteroids (> 8 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses are permitted in the absence of active autoimmune disease
* Known history of a positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS); HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dabrafenib and trametinib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* History of allergy or adverse drug reaction to the study drug components (nivolumab, dabrafenib, or trametinib) or drugs of similar chemical or biologic composition; patients with a history of severe hypersensitivity reaction to any monoclonal antibody should also be excluded
* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Uncontrolled intercurrent illness (requiring IV antibiotic treatment) including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and/or breastfeeding women are excluded from this study; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab, dabrafenib, and trametinib, breastfeeding should be discontinued if the mother is treated with nivolumab, dabrafenib, and trametinib; these potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2027-12-08 (Estimated); Study Completion 2027-12-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) as measured by Response Evaluation Criteria in Solid Tumors version 1.1 on both arms | From the time of initial response until documented tumor progression, assessed up to 3 years
  The ORR for each treatment group will be computed along 95% credible intervals.

SECONDARY OUTCOMES:
Incidence of adverse events assessed using National Cancer Institute's Common Terminology Criteria for Adverse Events version 4.0 | Up to 3 years
  The maximum grade of toxicity for each category of interest will be recorded for each patient and the summary results will be tabulated by category and grade. Will describe all dose limiting toxicities and other serious (>= grade 3) on a patient-by-patient basis; descriptions will include dose level and any relevant baseline data. Statistics on the number of cycles received by patients and any dose reductions will be tabulated.
Complete response | Up to 3 years
  Will be tabulated by disease diagnosis and by dose level; no formal statistical analyses are planned.
Partial response | Up to 3 years
  Will be tabulated by disease diagnosis and by dose level; no formal statistical analyses are planned.
Incidence of stable disease | From the start of the treatment until the criteria for progression are met, assessed up to 3 years
  Will be tabulated by disease diagnosis and by dose level; no formal statistical analyses are planned.
Overall survival (OS) | From treatment start date to last known vital sign, assessed up to 3 years
  The Kaplan-Meier method will be used to estimate OS. Associations between OS and clinical measures of interest will be determined using Cox proportional hazards regression models.
Progression-free survival (PFS) | From treatment start date to date of disease progression or death or the last evaluation date, assessed up to 3 years
  The Kaplan-Meier method will be used to estimate PFS. Associations between PFS and clinical measures of interest will be determined using Cox proportional hazards regression models.

OTHER OUTCOMES:
Circulating and tumor markers | Baseline up to 3 years
  Will be compared by the Wilcoxon signed-rank test. The false discovery rate will be controlled at 20% by the procedure of Benjamini and Hochberg's method.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein A Tawbi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org